CLINICAL TRIAL: NCT02515526
Title: Effect of Acute Ethanol Consumption on The Activity of Major Cytochrome P450 Enzymes, NAT2 and P-glycoprotein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Uwe Fuhr, Prof. Dr. Uwe Fuhr, University of Cologne
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EtOH_CYP_2013_KPUK
Record Dates: First submitted 2015-08-01; First posted 2015-08-04 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: AOD Effects and Consequences
MeSH Terms: interventions — Caffeine; Tolbutamide; Omeprazole; Dextromethorphan; Digoxin; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reference (Active Comparator): A cocktail of six different test substances to be administered orally followed by an I.V. dose of midzolam
  Interventions: Drug: caffeine, tolbutamide, omeprazole, dextromethorphan, digoxin, midazolam single doses
- Test (Experimental): A cocktail of six different test substances to be administered orally followed by an I.V. dose of midzolam. In addition, ethanol will be administered at six different time points with of reaching a blood alcohol concentration of 1 per mille to see its effect on the activity of major cytochrome P450 enzymes, NAT-2 and P-glycoprotein.
  Interventions: Drug: ethanol multiple doses plus caffeine, tolbutamide, omeprazole, dextromethorphan, digoxin, midazolam single doses

INTERVENTIONS:
Drug: caffeine, tolbutamide, omeprazole, dextromethorphan, digoxin, midazolam single doses — Reference period
  Other Names: Percoffedrinol, Tolbutamide PCH, Omepazol Ratiopharm, Hustenstiller Ratiopharm, Digacin and Midazolam-ratiopharm
  Arms: Reference
Drug: ethanol multiple doses plus caffeine, tolbutamide, omeprazole, dextromethorphan, digoxin, midazolam single doses — Test period
  Other Names: Percoffedrinol, Tolbutamide PCH, Omepazol Ratiopharm, Hustenstiller Ratiopharm, Digacin, Midazolam-ratiopharm and Wodka Gorbatschow 50%
  Arms: Test

SUMMARY:
Protocol title: Effect of acute alcohol consumption on the activity of major cytochrome P450 enzymes, NAT2 and P-glycoprotein.

Objectives: The study is mainly conducted to evaluate the effect of acute alcohol consumption on the activity of the most important drug metabolising cytochrome P450 enzymes CYP1A2, CYP2C9, CYP2C19, CYP2D6, intestinal CYP3A4, hepatic CYP3A4, NAT2 and on the activity of the drug transporter p-glycoprotein (intestinal and renal).

The study should also provide basis for a planned clinical study on interactions caused by chronic alcohol intake.

Design: Single center, open-label, two-way, cross-over study with randomly allocated sequences Test-Reference or Reference-Test.

The study is not a clinical drug study according to the German Drug Act.

Clinical phase: Not applicable

Volunteers: 16 healthy male and female subjects are planned for completion in accordance with the protocol, i.e. with evaluable/analysable data for all periods and treatments.

Clinical centre: Department of Pharmacology, Clinical Pharmacology Unit (KPH), University of Cologne, Gleueler Str. 24, 50931Köln, Germany

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Age: 18-55 years
* Normal body weight: (body mass index 18.5-30 kg/m2)
* Considered to be healthy on the basis of extensive pre-study screening
* Willing and capable to confirm written consent prior to enrolment after ample information has been provided.
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant ("clinically healthy"). The inclusion criterion "clinically healthy" will be determined both by physical examination and clinical-chemical tests which will be done prior to the clinical part of the study

Exclusion Criteria:

* subjects with any relevant clinical abnormality (as based on extensive medical history, physical examination, vital signs and 12-lead ECG)
* subjects with electrolyte disturbances
* subjects with any cardiac arrhythmia
* subjects with a history or evidence of hypertrophic obstructive cardiomyopathy
* subjects with a history or evidence of stenosis of the gastrointestinal tract
* subjects a history or evidence of ulcerative colitis
* subjects a history or evidence of toxic mega colon
* subjects with a history or evidence of myasthenia gravis
* subjects with evidence of chronic infections
* subjects with a history or evidence of bronchial asthma, COPD, pneumonia or other relevant respiratory diseases
* subjects with acute infections within the last two weeks
* subjects with a history of any allergic disease with clinical signs including hay fever and drug allergies
* subjects with suspicion of hypersensitivity to the investigational medications and/or subjects with a history of severe skin reactions
* subjects with any clinically relevant laboratory abnormality (incl. positive results for hepatitis and HIV serology)
* subjects receiving any medication within 1 week prior to study start or during the study (exceptions possible upon decision of Principal Investigator, e.g. paracetamol single dose for acute pain or topical acyclovir for herpes labialis)
* subjects who have taken a drug with a long half-life (> 24 hours) within four weeks before the first trial day
* subjects who received chronic drug treatment (> 3 days) within eight weeks before the first trial day
* subjects who participated in a trial with novel investigational medications within the last 8 weeks before the start of the present study
* subjects who participated in a trial with a registered compound within the last 4 weeks before the start of the present study
* subjects who donated blood or plasma within the last 4 weeks before the start of the present study
* actual smokers defined as subjects who smoked any cigarette during the last three months
* subjects who are known or suspected to be (social) drug dependent, incl. those drinking more than 50 g alcohol per day, those subjects must reduce their consumption to 30 g.
* subjects with a history of alcohol or recreational drug addiction
* subjects with positive drug screening tests
* subjects with a history of any severe disease that might interfere with the study objectives
* subjects who are not willing or able to abstain from alcohol, other than given as a study medication in the Reference period, methylxanthine-containing beverages and foods, caffeine containing products, papaver containing products and grapefruit flesh / juice starting from 72 hours before admission to the ward for the study until after the post screening tests
* subjects who adhere to a special diet (e.g. vegetarians) or lifestyle (incl. working at night and extreme physical activities such as competitive sports and weight lifting) that might interfere with the investigation
* subjects planning elective hospital treatment within one month after last intake of trial medication
* subjects who are known or suspected not to comply with the study directives and/or known or suspected not to be reliable or trustworthy
* subjects who are known or suspected not to be capable of understanding and evaluating the information that is given to them as part of the formal information policy (informed consent), in particular regarding the foreseeable risks and discomfort to which they will be exposed.
* Anticipated problems of successfully placing an indwelling venous catheter at the forearms

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
CYP1A2: AUC0-t of caffeine in plasma | 2 months
NAT2 activity: (AFMU + AAMU) / (AFMU + AAMU + 1X + 1U) | 2 months
CYP2C9: AUC0-t of tolbutamide in plasma | 2 months
CYP2C19: Molar omeprazole / 5-OH-omepazole AUC0-t ratio | 2 months
CYP2D6: Molar dextromethorphan / dextrorphan AUC0-t ratio | 2 months
Hepatic CYP3A4: hepatic clearance of midazolam | 2 months
Intestinal CYP3A4: intestinal extraction of midazolam | 2 months
Intestinal p-glycoprotein: absolute bioavailability of digoxin (calculated as Ae) | 2 months
Renal p-glycoprotein: renal secretion of digoxin | 2 months

SECONDARY OUTCOMES:
CYP1A2: Molar paraxanthine /caffeine AUC0-t ratio | 2 months
CYP2C9: Tolbutamide plasma concentration 24 h post-dose | 2 months
CYP2C19: AUC0-t of omeprazole in plasma | 2 months
CYP2C19: Molar omeprazole / 5-OH-omepazole plasma concentration ratio | 2 months
CYP2D6: AUC0-t of dextromethorphan in plasma | 2 months
CYP2D6: Molar dextromethorphan / dextrorphan plasma concentration ratio | 2 months
Intestinal p-glycoprotein: digoxin Cmax | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Fuhr, Principal Investigator — Department of Pharmacology,University Hospital Cologne
Locations (1):
- Department of Pharmacology I, University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Hsin CH, Stoffel MS, Gazzaz M, Schaeffeler E, Schwab M, Fuhr U, Taubert M. Combinations of common SNPs of the transporter gene ABCB1 influence apparent bioavailability, but not renal elimination of oral digoxin. Sci Rep. 2020 Jul 27;10(1):12457. doi: 10.1038/s41598-020-69326-y. PMID 32719417